CLINICAL TRIAL: NCT00495638
Title: Pulmonary Hypertension and the Hypoxic Response in SCD
Brief Title: Pulmonary Hypertension, Hypoxia and Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070181; 07-H-0181
Record Dates: First submitted 2007-06-30; First posted 2007-07-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-12-02

CONDITIONS: Chuvash Polycythemia; Cerebrovascular Disease; Pulmonary Hypertension; Sickle Cell Anemia
Keywords: 6-Minute Walk; Chuvash Polycythemia; Echocardiogram; Sickle Cell Anemia; Pulmonary Function Tests; Sickle Cell Disease; SCD; Pulmonary Hypertension
MeSH Terms: conditions — Cerebrovascular Disorders; Hypertension, Pulmonary; Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The study will look at the risk factors for pulmonary hypertension (high blood pressure in the lungs) in children and adolescents with sickle cell anemia (SCA) and examine the role of hypoxia (oxygen shortage) in the disease. In patients with SCA, red blood cells become sickle-shaped and tend to form clumps that get stuck in blood vessels, blocking blood flow to the limbs and organs. Blocked blood vessels can cause pain, serious infections, and organ damage. Many patients with SCA also develop pulmonary hypertension.

Children and adolescents with SCA or Chuvash polycythemia (another blood disorder that carries an increased risk for pulmonary hypertension) may be eligible for this study.

Participants undergo the following procedures at the beginning (baseline) and end of the study:

* History, physical examination and blood tests .
* Echocardiography (ultrasound study of heart function).
* Transcranial doppler (brain ultrasound study to measure brain blood flow).
* Lung function tests.
* 6-minute walk (measure of the distance covered in 6 minutes of walking).

In addition, patients are followed by telephone or by clinic visits every 6 months for a review of their medical history and medications. A physical examination is also done at 12 months.

DETAILED DESCRIPTION:
The research is designed to determine the prevalence and risk factors of pulmonary hypertension (PHT) in children and adolescents with sickle cell disease (SCD), and to determine the role of the hypoxic response in its pathogenesis. In this regard, proliferative vascular responses mediated by (i) hypoxia inducible factor (HIF)-regulated pathways and (ii) nitric oxide (NO)-scavenging will be compared between patients with SCD and patients with Chuvash polycythemia (CP), another hematological disorder characterized by increased risk for PHT. High throughput microarray and genotyping technologies will be employed to identify candidate gene pholymorphisms involved in pathologic responses to hypoxia in SCD and CP patients with and without PHT.

ELIGIBILITY:
* INCLUSION CRITERIA

A. For PAH in children and adolescents with SCD:

Inclusion criteria for all participants:

1. The informed consent has been signed by the participant, parent or legal guardian as appropriate.
2. Age of 3 to 20 years.

Inclusion criteria for SCD patients:

1. Diagnosis of sickle cell disease (electrophoretic HPLC documentation of SS, SC, Sb thalassemia or other major sickling phenotype such as SD, SO-Arab or SLepore is required).
2. At least three weeks has elapsed since hospitalization for acute chest syndrome, pain crisis, infection or other complication of SCD.
3. Absence of acute infection, pain crisis, or other acute complication of SCD. (Chronic SCD complications such as stuttering priapism, stable chronic pain and leg ulcers are not reasons for exclusion.)

Inclusion criteria for control participants:

1. Self-described race is African American.
2. Absence of diagnosis of SCD as defined above and subsequent electrophoretic or HPLC documentation.
3. Absence of acute infection, injury, surgery or asthmatic episode.

EXCLUSION CRITERIA:

Exclusion criteria for all participants:

1. Age of less than 3 years or 21 years or more at time of enrollment.
2. Presence of acute infection, pain crisis, injury, surgery, asthmatic episode or other acute complication.

Exclusion criteria for SCD patients:

1. Hemoglobin A only phenotype, hemoglobin S trait or hemoglobin C trait.
2. Less than three weeks has elapsed since hospitalization for acute chest syndrome, pain crisis, infection or other complication of SCD.

Exclusion criteria for control participants:

1. Self-described ethnicity other than African American.
2. Diagnosis of SCD or electrophoretic or HPLC documentation of major sickling phenotype as described above.

B. Angiogenic and vasomotor responses mediated by HIF-regulated pathways in patients with SCD and CP with and without PAH.

INCLUSION CRITERIA:

Inclusion criteria for all participants:

1. The informed consent has been signed by the participant, parent or legal guardian as appropriate.
2. Age of 3 years or greater.
3. Absence of acute infection, pain crisis, cerebral vascular accident, thrombosis or other acute complication.

Inclusion criteria for SCD or CP patients with PAH:

1. Diagnosis of SCD and electrophoretic or HPLC documentation of SS, SC, Sbeta thalassemia or other major sickling phenotype such as SD, SO-Arab or SLepore OR diagnosis of CP and evidence of homozygosity for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine.
2. At least three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV of 2.5 m/sec or greater.

Inclusion criteria for SCD or CP patients without PAH:

1. Diagnosis of SCD and electrophoretic or HPLC documentation of SS, SC, Sb thalassemia or other major sickling phenotype such as SD, SO-Arab or SLepore OR diagnosis of CP and evidence of homozygosity for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine.
2. At least three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV less than 2.5 m/sec.
4. Matched by age (plus or minus 2 years), sex and ethnicity to a specific patient with SCD and PAH or CP and PAH enrolled for this same study.

Inclusion criteria for control participants:

1. Absence of diagnosis of SCD as defined above and subsequent electrophoretic documentation.
2. Absence of diagnosis of CP and subsequent documentation of VHL 598 wildtype.
3. At least three weeks has elapsed since hospitalization for illness or surgery.
4. Matched by age (plus or minus 2 years) and sex and ethnicity to a specific patient with SCD and PAH or CP and PAH enrolled for this same study.
5. Absence of diagnosis of PAH, anemia, or polycythemia.

EXCLUSION CRITERIA:

Exclusion criteria for all participants:

1. Age of less than 3 years.
2. Presence of a condition associated with secondary PAH other than SCD or CP, such as collagen vascular disease, congenital heart disease, or chronic lung disease.
3. Presence of acute infection, injury, surgery, asthmatic episode, pain crisis, cerebral vascular accident, thrombosis or other acute complication.

Exclusion criteria for SCD or CP patients with PAH:

1. Hemoglobin AA only phenotype, hemoglobin S trait, hemoglobin C trait for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine heterozygosity or VHL wildtype.
2. Less than three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV less than 2.5 m/sec.

Exclusion criteria for SCD or CP patients without PAH:

1. Hemoglobin AA only phenotype, hemoglobin S trait, hemoglobin C trait OR for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine heterozygosity or VHL wildtype.
2. Less than three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV greater than or equal to 2.5 m/sec.

Exclusion criteria for control participants:

1. Diagnosis of SCD or electrophoretic or HPLC evidence of major sickling phenotype as described above OR diagnosis of CP or for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine homozygosity.
2. ECHO-determined TRV greater than or equal to 2.5 m/sec.

C. High throughput microarray and genotyping technologies to identify candidate gene polymorphisms involved in pathologic responses to hypoxia in SCD and CP patients with PAH.

INCLUSION CRITERIA:

Inclusion criteria for all participants:

1. The informed consent has been signed by the participant, parent or legal guardian as appropriate.
2. Age of 3 years or greater.
3. Absence of acute infection, pain crisis, cerebral vascular accident, thrombosis or other acute complication.

Inclusion criteria for SCD or CP patients with PAH:

1. Diagnosis of SCD and electrophoretic or HPLC documentation of SS, SC, Sb thalassemia or other major sickling phenotype such as SD, SO-Arab or SLepore OR diagnosis of CP and evidence of homozygosity for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine.
2. At least three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV of 2.5 m/sec or greater.

Inclusion criteria for SCD or CP patients without PAH:

1. Diagnosis of SCD and electrophoretic or HPLC documentation of SS, SC, Sb thalassemia or other major sickling phenotype such as SD, SO-Arab or SLepore OR diagnosis of CP and evidence of homozygosity for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine.
2. At least three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
3. ECHO-determined TRV less than 2.5 m/sec
4. Matched by age (plus or minus 2 years), sex and ethnicity to a specific patient with SCD and PAH or CP and PAH enrolled for this same study.

Inclusion criteria for screening for population prevalence of polymorphisms:

1. Absence of diagnosis of SCD, CP or PAH.
2. Self-described African-American or Chuvash ethnicity.

EXCLUSION CRITERIA:

Exclusion criteria for all participants:

1. Age of less than 3 years.
2. Presence of acute infection, injury, surgery, asthmatic episode, pain crisis, cerebral vascular accident, thrombosis or other acute complication.

Exclusion criteria for SCD or CP patients with PAH:

1. Hemoglobin AA only phenotype, hemoglobin S trait, hemoglobin C trait OR for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine heterozygosity or VHL wildtype.
2. Presence of a condition associated with secondary PAH other than SCD or CP, such as collagen vascular disease, congenital heart disease, or chronic lung disease.
3. Less than three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
4. ECHO-determined TRV less than 2.5 m/sec.

Exclusion criteria for SCD or CP patients without PAH:

1. Hemoglobin AA only phenotype, hemoglobin S trait, hemoglobin C trait OR for mutation of the von Hippel-Lindau gene at position 598 from cytosine to thymidine heterozygosity or VHL wildtype.
2. Presence of a condition associated with secondary PAH other than SCD or CP, such as collagen vascular disease, congenital heart disease, or chronic lung disease.
3. Less than three weeks has elapsed since hospitalization for SCD (acute chest syndrome, pain crisis, infection or other complication) or CP (cerebral vascular accident, thrombotic event or other complication).
4. ECHO-determined TRV greater than or equal to 2.5 m/sec.

Exclusion criteria for screening for population prevalence of polymorphisms

1. Diagnosis of SCD, CP or PAH.
2. Self-described ethnicity other than African-American or Chuvash.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06-28; Study Completion 2014-12-02

CONTACTS AND LOCATIONS:
Overall Officials: Caterina P Minniti, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (7):
- United States (6):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Baylor College of Medicine, Houston, Texas
- Republic Cardiac Center in Cheboksary, Chuvashia, Russia

REFERENCES:
- [Derived] Sable CA, Aliyu ZY, Dham N, Nouraie M, Sachdev V, Sidenko S, Miasnikova GY, Polyakova LA, Sergueeva AI, Okhotin DJ, Bushuev V, Remaley AT, Niu X, Castro OL, Gladwin MT, Kato GJ, Prchal JT, Gordeuk VR. Pulmonary artery pressure and iron deficiency in patients with upregulation of hypoxia sensing due to homozygous VHL(R200W) mutation (Chuvash polycythemia). Haematologica. 2012 Feb;97(2):193-200. doi: 10.3324/haematol.2011.051839. Epub 2011 Oct 11. PMID 21993671
- [Derived] Darbari DS, Onyekwere O, Nouraie M, Minniti CP, Luchtman-Jones L, Rana S, Sable C, Ensing G, Dham N, Campbell A, Arteta M, Gladwin MT, Castro O, Taylor JG 6th, Kato GJ, Gordeuk V. Markers of severe vaso-occlusive painful episode frequency in children and adolescents with sickle cell anemia. J Pediatr. 2012 Feb;160(2):286-90. doi: 10.1016/j.jpeds.2011.07.018. Epub 2011 Sep 3. PMID 21890147